CLINICAL TRIAL: NCT04925271
Title: Closure of Mucosal and Submucosal Defects in the Gastrointestinal Tract Using the Novel X-Tack Endoscopic Suturing Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Anand Kumar, Associate Professor of Medicine, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21D.166
Record Dates: First submitted 2021-05-31; First posted 2021-06-14 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Polyp of Colon; Fistula
Keywords: Endoscopic submucosal dissection; Suturing
MeSH Terms: conditions — Colonic Polyps; Fistula

STUDY DESIGN:
Intervention Model Description: Patients undergoing closure of a mucosal or submucosal defect in the gastrointestinal tract will be randomized 1:1 to either closure with X-Tack or closure with Overstitch.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- X-Tack (Experimental): The gastrointestinal tract mucosal or submucosal defect is closed using the X-Tack device.
  Interventions: Device: X-Tack
- Overstitch (Active Comparator): The gastrointestinal tract mucosal or submucosal defect is closed using the Overstitch device.
  Interventions: Device: Overstitch

INTERVENTIONS:
Device: X-Tack — The mucosal or submucosal defect is closed with X-Tack.
  Arms: X-Tack
Device: Overstitch — The mucosal or submucosal defect is closed with Overstitch.
  Arms: Overstitch

SUMMARY:
After removing large polyps from the gastrointestinal tract, gastroenterologists close the new defect with devices to prevent complications like bleeding or the development of a leak. Commonly, this is done with a device called Overstitch, which allows the gastroenterologist to stitch the defect with an endoscope. A new device called X-tack has been developed to simplify endoscopic stitching. In this study, the new X-tack device will be compared to Overstitch when closing defects in the gastrointestinal tract. The two devices will be compared to see how long it takes to close a defect, as well as if there are any differences in complications like bleeding or infection.

DETAILED DESCRIPTION:
Currently, the community standard is that gastroenterologists who are familiar with Overstitch start using the X-Tack without additional training. However, a hands-on demonstration session with the X-Tack device in a "dry lab" has been conducted with each endoscopist in the trial prior to the study in order to familiarize them with device before enrollment. Each endoscopist has also participated in a "wet lab" using an explant (porcine stomach) to simulate in vivo closure of defects using the X-Tack system. The device operates in a similar fashion compared to previous suturing devices, which are used frequently by all endoscopists involved in this study. On this basis, all endoscopists in the study report comfort and familiarity with the X-Tack system, and the "break-in" period is not anticipated to affect safety or results during the study. The primary study visit will be comprised of the endoscopic procedure at the time of defect closure and a telephone call 48-72 hours later to assess for complications. Patient will be enrolled in the pre-procedure area. If the patient has a pre-procedure visit, they may be notified of their potential for enrollment in the study at that time, though not all patients have a pre-procedure visit in our practice. Patients will be randomized to closure with the X-Tack system versus closure with the Overstitch system prior to their procedure using a centralized computer-generated randomization. Technical success of closure, time of closure, number of sutures required, need for alternative modalities for closure, and any intraprocedural complications (bleeding, perforation) will be recorded. Any patient with possible periprocedural perforation will receive antibiotics at the endoscopist's discretion. At the endoscopist's discretion, the patient may cross over during the procedure to the other group if they believe that their current closure strategy is failing to safely close the defect. Alternate methods of closure (TTS clips, over-the-scope clips) may be used in either group if required by the endoscopist for safe closure of the defect. After the procedure, most patients are observed in the recovery area for 1-2 hours for any signs of complications before they are discharged home.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Undergoing closure of a gastrointestinal luminal defect for which a suturing device would be otherwise indicated

Exclusion Criteria:

* INR > 2
* Platelets < 150
* Ongoing anticoagulation not meeting ASGE Antithrombotic Guidelines (Acosta RD et al, The Management of Antithrombotic Agents for Patients Undergoing GI Endoscopy, Gastrointest Endosc, 2016; 83(1): 3-16)
* Hemodynamic instability
* Ongoing or anticipated pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Kumar, MD MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any publications from the trial after deidentification (text, tables, figures and appendices) will be made available upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication, no end date.
Access Criteria: Proposals should be directed to anand.kumar@jefferson.edu.

REFERENCES:
- [Background] Kothari ST, Huang RJ, Shaukat A, Agrawal D, Buxbaum JL, Abbas Fehmi SM, Fishman DS, Gurudu SR, Khashab MA, Jamil LH, Jue TL, Law JK, Lee JK, Naveed M, Qumseya BJ, Sawhney MS, Thosani N, Yang J, DeWitt JM, Wani S; ASGE Standards of Practice Committee Chair. ASGE review of adverse events in colonoscopy. Gastrointest Endosc. 2019 Dec;90(6):863-876.e33. doi: 10.1016/j.gie.2019.07.033. Epub 2019 Sep 25. PMID 31563271
- [Background] Pohl H, Grimm IS, Moyer MT, Hasan MK, Pleskow D, Elmunzer BJ, Khashab MA, Sanaei O, Al-Kawas FH, Gordon SR, Mathew A, Levenick JM, Aslanian HR, Antaki F, von Renteln D, Crockett SD, Rastogi A, Gill JA, Law RJ, Elias PA, Pellise M, Wallace MB, Mackenzie TA, Rex DK. Clip Closure Prevents Bleeding After Endoscopic Resection of Large Colon Polyps in a Randomized Trial. Gastroenterology. 2019 Oct;157(4):977-984.e3. doi: 10.1053/j.gastro.2019.03.019. Epub 2019 Mar 15. PMID 30885778
- [Background] Qumseya BJ, Wolfsen C, Wang Y, Othman M, Raimondo M, Bouras E, Wolfsen H, Wallace MB, Woodward T. Factors associated with increased bleeding post-endoscopic mucosal resection. J Dig Dis. 2013 Mar;14(3):140-6. doi: 10.1111/1751-2980.12002. PMID 23134152
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Kantsevoy SV, Bitner M, Mitrakov AA, Thuluvath PJ. Endoscopic suturing closure of large mucosal defects after endoscopic submucosal dissection is technically feasible, fast, and eliminates the need for hospitalization (with videos). Gastrointest Endosc. 2014 Mar;79(3):503-7. doi: 10.1016/j.gie.2013.10.051. Epub 2013 Dec 12. PMID 24332082
- [Background] Zhang QS, Han B, Xu JH, Gao P, Shen YC. Clip closure of defect after endoscopic resection in patients with larger colorectal tumors decreased the adverse events. Gastrointest Endosc. 2015 Nov;82(5):904-9. doi: 10.1016/j.gie.2015.04.005. Epub 2015 May 12. PMID 25975527
- [Background] ASGE Standards of Practice Committee; Acosta RD, Abraham NS, Chandrasekhara V, Chathadi KV, Early DS, Eloubeidi MA, Evans JA, Faulx AL, Fisher DA, Fonkalsrud L, Hwang JH, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Shaukat A, Shergill AK, Wang A, Cash BD, DeWitt JM. The management of antithrombotic agents for patients undergoing GI endoscopy. Gastrointest Endosc. 2016 Jan;83(1):3-16. doi: 10.1016/j.gie.2015.09.035. Epub 2015 Nov 24. No abstract available. PMID 26621548
- [Derived] Agnihotri A, Mitsuhashi S, Holmes I, Kamal F, Chiang A, Loren DE, Kowalski TE, Schlachterman A, Kumar AR. Randomized trial of gastric and colorectal endoscopic submucosal dissection defect closure comparing a novel through-the-scope suturing system with an over-the-scope suturing system (with video). Gastrointest Endosc. 2024 Feb;99(2):237-244.e1. doi: 10.1016/j.gie.2023.07.046. Epub 2023 Aug 1. PMID 37536633

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | X-Tack | Overstitch
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | X-Tack | Overstitch | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 61.8 (13.5) | 62.2 (12.2) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 14 | 16 | 30
  Race/Ethnicity: Black | 4 | 1 | 5
  Race/Ethnicity: Asian | 2 | 2 | 4
  Race/Ethnicity: Hispanic | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Closure
Description: The time required to close the defect using the device
Time Frame: At time of endoscopy
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | X-Tack | Overstitch
Number analyzed (Participants) | 20 | 20
minutes | 23.3 (13.9) | 18.4 (16.9)

2. Secondary Outcome: Incomplete Closure
Description: Either crossover to the other study group per endoscopist's discretion, or the need for additional modalities to close the defect such as endoscopic clips
Time Frame: At time of endoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | X-Tack | Overstitch
Number analyzed (Participants) | 20 | 20
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | X-Tack | Overstitch
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | X-Tack (N=20) | Overstitch (N=20)
Delayed bleeding (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT04925271/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT04925271/ICF_001.pdf